CLINICAL TRIAL: NCT02099877
Title: Observational Study: The Effect of μ-opioid Receptor Genetic Polymorphism on Neuraxial Opioid Labor Analgesia
Brief Title: μ-opioid Receptor Polymorphism and Opioid Analgesia
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sahar Sayyid, Professor, American University of Beirut Medical Center
Other Study IDs: ANES.SS.11
Record Dates: First submitted 2014-03-25; First posted 2014-03-31 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Pharmacogenetic and Duration of Labor Fentanyl Analgesia
Keywords: µ-opioid receptor polymorphism; Opioids; Opioid analgesia; Labor analgesia
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nulliparous requesting epidural: Nulliparous parturients ≥ 37 weeks gestation, with ASA I or II, with an uncomplicated course of singleton vertex pregnancy requesting epidural analgesia for pain relief will be included.
  When the patient requests analgesia, cervical dilatation will be verified by the obstetric resident/attending. Then epidural analgesia will be initiated with a test dose of 3mL of 2% lidocaine and epinephrine 15 µg and a dose of fentanyl 100 µg diluted to a total volume of 10 mL with preservative- free normal saline. Before placement of the epidural, venous blood (2 mL) will be drawn into special tubes. Genotyping of OPRM1: p.118A/G will be also performed.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Epidural analgesia will be initiated with 100µg of epidural fentanyl

SUMMARY:
In this prospective observational double-blind study, the investigators aim to assess the effect of the single nucleotide polymorphism of the μ-opioid receptor gene (OPRM1, p.118A/G) on the duration of epidural fentanyl labor analgesia.

DETAILED DESCRIPTION:
The single nucleotide polymorphism (SNP), p.118A/G of the µ -opioid receptor gene (OPRM1), may alter pain perception and individual response to opioid analgesia. This SNP leads to a variant µ-opioid receptor in which an asparagine is substituted for aspartate as the 102nd amino acid of the receptor protein (p.Asn102Asp). At the investigators' institution, it is common practice to initiate labor analgesia with epidural fentanyl. No data are available to determine how the µ-opioid polymorphism affects pain perception and response to opioids, such as fentanyl, in the investigators' population. The investigators aim to assess the effect of the single nucleotide polymorphism of the µ-opioid receptor gene (OPRM1, p.118A/G) on duration of epidural fentanyl labor analgesia.

This is a prospective observational and double-blind study. Before initiation of epidural labor analgesia, venous blood will be drawn into coded EDTA tubes. DNA isolation and genotyping of OPRM1:p.118A/G will be performed at the American University of Beirut. In 250 parturients, labor epidural analgesia will be initiated with 100 µg of epidural fentanyl following a test dose of lidocaine and epinephrine. No drugs will be injected until second request of analgesia. Patients will be divided into two groups based on their genetic groups: Group A consists of wild-type homozygote (A118), and Group G includes heterozygote and homozygote carrying the G118 allele. Duration of fentanyl analgesia (primary outcome) will be compared. Data will be presented as a mean ± SD or numbers and percentages. Statistical analysis will be performed with the Student's t-test, Chi-square or Fisher's exact test as appropriate. P value <0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous parturients ≥ 37 weeks gestation, with ASA I or II, with an uncomplicated course of singleton vertex pregnancy (in spontaneous labor or with spontaneous rupture of membrane), requesting epidural analgesia for pain relief

Exclusion Criteria:

* Advanced cervical dilation (> 5 cm) at the time of request for epidural analgesia
* Severe medical or obstetric complications (preeclampsia, uncontrolled pregestational diabetes, etc…)
* Multiple gestation
* Contraindication to epidural analgesia
* Local anesthetics or fentanyl allergy
* History of chronic opioid use or recent acute opioid use.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous parturients ≥ 37 weeks gestation, with ASA I or II, with an uncomplicated course of singleton vertex pregnancy requesting epidural analgesia for pain relief
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Duration of epidural fentanyl | up to 24h
  The primary outcome variable is duration of epidural fentanyl for labor analgesia.

SECONDARY OUTCOMES:
VAS at request for analgesia | up to 24h
Cervical dilation at request for analgesia | up to 24h
Incidence of pruritus, nausea, and vomiting. | up to 24h

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Siddik Sayyid, MD, Principal Investigator — American Univesity of Beirut
Locations (1):
- American University of Beirut, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No